CLINICAL TRIAL: NCT03111225
Title: Thoracic Paraspinal Soft Tissue Mobilizations in Treatment of Patients With Upper Limb Complex Regional Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reuth Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Reuth Research Institute, Professor, Reuth Rehabilitation Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-2
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Complex Regional Pain Syndromes
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Intervention Model Description: The observation stage is a case- control study, the treatment stage is an A-B-A design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRPS patients (Experimental): CRPS patients that will be examined for trigger points in the thoracic muscles. 10 out of the 23 will also be included in the intervention stage and will recieve a month of conventional physiotherapy, and a month of conventional physiotherapy with addition of massage to the thoracic area.
  Interventions: Diagnostic Test: massage
- healthy controls (No Intervention): healthy controls that will be examined for trigger points in the thoracic muscles (and will be compared to the CRPS patients)

INTERVENTIONS:
Diagnostic Test: massage — a 15 minutes thoracic massage will be added to the regular physical therapy treatment
  Arms: CRPS patients

SUMMARY:
This study examines the prevalence of trigger points in muscles in the thorax in upper limb Complex Regional Pain Syndrome (CRPS) patients, compared to healthy subjects. In addition, we will examine if adding treatment to muscles in the thoracic area (to the regular physical therapy treatment) will alleviate some of the sensitivity in the upper limb in CRPS patients.

DETAILED DESCRIPTION:
This study examines the prevalence of trigger points in muscles in the thorax in upper limb Complex Regional Pain Syndrome (CRPS) patients, compared to healthy subjects. The muscles that will be examined are: Subclavius, Pectoralis minor, Rhomboids, Infraspinatus and Serratus superior posterior.

In addition, we will examine if adding treatment to muscles in the thoracic area (to the regular physical therapy treatment) will alleviate some of the sensitivity in the upper limb in CRPS patients.This will be examined in an A-B-A design: at first the patients will be examined. Then they will recieve conventional physiotherapy treatment for a month. After a month, they will be examined again, and then they will recieve soft tissue massage to the thoracic area for 15 minutes in addition to the conventional physiotherapy treatment. After a month of the combined treatment, the patients will be examined a third and final time.

ELIGIBILITY:
Inclusions Criteria for "cases" in stage 1 and all subjects of stage 2:

* Age between 18-70
* CRPS diagnosed by board certified specialist in rehabilitation or pain medicine
* Constant chronic pain for ≥six months preceding the trial;
* Spontaneous pain in a day of first evaluation (numeric pain rating scale (NPRS) ≥4/10)
* Stimulated pain is not attributable to other causes, such as peripheral inflammation.

Inclusions Criteria for "controls" in stage 1:

* Age between 18-70
* Do not suffer from any medical issues or chronic pain

Exclusion criteria for all subjects in stages 1 and 2:

* Tumors
* Participation in another interventional clinical trial.
* History of major psychiatric or neurological illness (like stroke).
* Rheumatoid arthritis or other major rheumatologic disorders.
* Fibromyalgia or any other systemic illness.
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | 10 minutes
  Questionnaire that examines upper limb function

SECONDARY OUTCOMES:
Goniometer | 1 minute
  shoulder flexion range of motion
CRPS severity score (CSS) | 20 minutes
  form filled by an MD after an interview and examination of a patient
skin rolling test | 1 minute
trigger point examination | 5 minutes
NPRS | 1 minute
  Numerical Pain Rating Scale
Pressure algometer | 10 minutes
  pressure pain threshold
Allodynia in scapula, arm and forearm | 5 minutes
  von Frey filaments

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jeaques Vatine, Prof, Principal Investigator — Reuth Rehabilitation Hospital
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No